CLINICAL TRIAL: NCT05521906
Title: Development and Pilot Evaluation of an Online Intervention to Prevent Dating Violence and Problem Drinking in Sexual Minority Youth
Brief Title: Evaluation of PRYSHM for LGBTQIA2S+ Youth
Acronym: PRYSHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: University of Houston (Other); University of Colorado, Colorado Springs (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21985IRB; R34AA028401 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Dating Violence; Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: SGMY (N=300) are randomly assigned to a treatment (n=200) or wait-list (n=100) control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Condition (Experimental): The PRYSHM program is theoretically grounded, follows best practices for effective health behavior prevention, and includes nine, one hour sessions co-facilitated by 2 LGBTQ+ adults.
  Interventions: Behavioral: Promoting Resilient Youth with Strong Hearts and Minds (PRYSHM)
- Control (No Intervention): Check-ins/provision of resources

INTERVENTIONS:
Behavioral: Promoting Resilient Youth with Strong Hearts and Minds (PRYSHM) — The intervention focuses on psycho-education (provision of accurate information about LGBTQIA2S+ people, education about the effects of alcohol), fostering positive identity development for LGBTQIA2S+ youth (e.g., fostering pride in identity, exposure to positive adult role models), teaching of alcohol use and sexual refusal skills, correction of inaccurate social norms about alcohol use and dating violence, teaching assertive communication skills, teaching emotion coping skills, mindfulness and grounding skills, and teaching bystander intervention skills related to dating/sexual violence and alcohol use..
  Arms: Treatment Condition

SUMMARY:
The overarching goal of the proposed project is to develop an innovative, online synchronous DV and AU prevention curriculum created specifically for SGMY (ages 15 to 18); conduct a pilot randomized controlled trial to assess its feasibility and acceptability of the intervention and study procedures; identify preliminary outcomes of the intervention; and ensure that the intervention is working equally well for SGMY of color.

DETAILED DESCRIPTION:
Alcohol use (AU) is strongly associated with dating violence (DV), and both DV and AU occur at alarmingly high rates among youth. Sexual and gender minority youth (SGMY) are no exception. Research suggests that DV and AU affects SGMY at rates significantly higher than cisgender heterosexual youth. This increased risk can be explained by experiences of minority stress, specifically distal stressors (e.g., discrimination experienced as a result of one's SOGIE [sexual orientation and gender identity and expression] status) and proximal stressors, including identity concealment (hiding one's SOGIE from others), and internalized homo/bi/transphobia (e.g., feeling ashamed of one's sexual orientation/gender identity, wishing one was not LGBTQ+). Whereas minority stress increases the risk for DV and AU, having a sense of community (e.g., sense of belonging, emotional connectedness) with other SGMY reduces the risk for DV and AU.

Prevention programming that targets proximal minority stressors and sense of community, in conjunction with evidence-based DV and AU prevention programming components (e.g., bystander intervention, refusal skills, correcting misperceptions of social norms, protective behavioral strategies), could reduce rates of DV and AU among SGMY. Also, because minority stress and sense of community are risk factors in the etiological pathways to other problematic health behaviors (e.g., sexual risk-taking), reducing minority stress, and increasing a sense of community among SGMY presumably may decrease other risk behaviors (e.g., drug use) and depressive symptoms. To date, however, no such programming exists for SGMY. In fact, DV and AU prevention programming has been widely criticized for lacking inclusive information for, as well as representations of, SGMY and universal DV programs do not work for SGMY. Further, although not specific to SGMY, universal DV programs do not work for youth of color, and SGMY of color experience the highest rates of DV and AU, underscoring the urgency for which DV and AU prevention programs for multiply minoritized SGMY, including those in hard to reach areas (e.g., rural communities), are needed.

Following a Stage 1A and 1B model, the proposed project seeks to develop and evaluate via a randomized controlled pilot study an online DV and AU prevention initiative for SGMY (15 to 18 years old), entitled Promoting Resilient Youth with Strong Hearts and Minds (PRYSHM). The PRYSHM program is theoretically grounded, follows best practices for effective health behavior prevention, and includes eight one hour sessions co-facilitated by two LGBTQIA2S+ adults. Use of synchronous online delivery via web-based teleconference was selected for PRYSHM given that a notable portion of SGMY are not out and thus may not have the opportunity to participate in an in-person program. This could be especially true for youth living in rural and remote areas of the U.S. where rates of minority stress are highest and sense of community is lowest (of note, the vast majority of youth in rural areas own smartphones). Also, research suggests that more than half of SGMY (both out and not-out youth) are members of an online LGBTQIA2S+ community, further underscoring the probable utility, scalability, and cost-effectiveness of online delivery of the PRYSHM.

Specific Aims of this R34 intervention development grant are as follows:

Aim 1: Development Phase: Finalize and refine PRYSHM materials through key informant feedback (i.e., SGMY advisory board, experts in the field) (Aim 1a) and conduct an open pilot trial with ten dating SGMY (Aim 1b).

Aim 2: Pilot Evaluation Phase: Recruit 300 dating SGMY via social media and other online advertisements and randomly assign them to a wait-list control condition (n = 100) or PRYSHM condition (n = 200) (Aim 2a). Assess acceptability and feasibility of the program and research procedures via post-session surveys, program observations, and online exit interviews with a subsample of youth (n = 20 or until saturation is achieved) (Aim 2b). Pre-, immediate, and 3-month posttests will be used to assess the acceptability of the study procedures (e.g., compliance with surveys) and generate initial data on the efficacy of PRYSHM in reducing DV and AU (Aim 2c). Exploratory analyses will examine mediators (e.g., sense of community, ethnic/racial cultural identity) and moderators (e.g., demographics [race/ethnicity, gender identity, dosage]) of treatment effects. Guided by intersectional literature that suggests not using comparative methods and sample size limitations, we will examine the treatment effects within groups of SGMY of color to determine promise of efficacy (Aim 2d).

This project is highly significant as it: (1) addresses DV and AU and related deleterious health behaviors (critical U.S. public health problems) among multiply minoritized SGMY; (2) can reach SGMY in rural and remote regions of the U.S. who experience the highest rates of minority stress and lowest sense of community; and (3) tests a scalable prevention strategy with the potential for paramount public health impact. This study is innovative as it is the first to test the effects of a group-based, online synchronous DV and AU prevention program tailored explicitly for diverse SGMY.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as LGBTQIA2S+ (sexual and/or gender minority), and/or report being unsure of their sexual orientation, and/or report experiencing romantic/sexual attraction to someone of the same sex assigned at birth.
* Age between 15 and 18 years.
* Ability to read and speak in English.
* Current residence in the United States.
* Consistent access to an electronic device (e.g., smartphone, tablet, computer) with high speed Internet access and/or Wi-Fi.
* Ability to attend 9 weekly, one hour online intervention sessions.
* Recent or currently in a dating/romantic/sexual relationship (past three months).
* Not at high risk for suicide (as defined by not endorsing a critical item on a past-month suicide screening measure [SBQ-R], and/or not be deemed at elevated risk for suicide on the basis of a clinical interview,)

Exclusion Criteria:

* Age under 15 or over 18 years.
* Identify as heterosexual and cisgender.
* Current enrollment as a full-time college student.
* Lack of English language proficiency (either written and/or spoken).
* Current residence outside of the U.S.
* No current or recent (in past three months) dating/romantic/sexual relationship.
* No consistent access to an electronic device (e.g., smartphone, tablet, computer) with high speed Internet or Wi-Fi.
* Inability to attend scheduled weekly one hour intervention sessions.
* Elevated risk of suicidality (reporting a past month suicide attempt or past month suicide threat with intent to die on the SBQ-R or determined to be at elevated current risk for suicidality based on a clinical interview).

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 314 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska (Lincoln), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD (using pseudoGUIDS) will be uploaded into the NIAAA data repository consistent with NIAAA policy for studies funded by NIAAA. The data in the NIAAA data archive are catalogued and made available to the general research community after a two year embargo period following the end date of the research award.
Time Frame: IPD will be available after a 2 year embargo period from the award end date. IPD will be available within the NIAAA data archive in perpetuity.
Access Criteria: To access to IPD from within the NIAAA data archive, researchers will need to receive authorization by completing the NDA Data Access Request (DAR) and satisfying several pre-requisites. DARs will be reviewed by a special committee at NIAAA to ensure that the researcher has made an adequate case for the responsible use of the data. Individuals seeking access to IPD must be associated with an NIH recognized institution with an FWA and must provide a research-related need to access the data.
URL: https://nda.nih.gov/niaaa/getting-data-access.html

REFERENCES:
- [Background] Edwards KM, Banyard VL, Sessarego SN. Dating and sexual violence victimization and perpetration among high school youth: Incidence and correlates. Manuscript in preparation. 2017.
- [Background] Edwards KM. Incidence and Outcomes of Dating Violence Victimization Among High School Youth: The Role of Gender and Sexual Orientation. J Interpers Violence. 2018 May;33(9):1472-1490. doi: 10.1177/0886260515618943. Epub 2015 Dec 13. PMID 26668180
- [Background] Vagi KJ, O'Malley Olsen E, Basile KC, Vivolo-Kantor AM. Teen Dating Violence (Physical and Sexual) Among US High School Students: Findings From the 2013 National Youth Risk Behavior Survey. JAMA Pediatr. 2015 May;169(5):474-82. doi: 10.1001/jamapediatrics.2014.3577. PMID 25730143
- [Background] Baiocco R, D'Alessio M, Laghi F. Binge drinking among gay, and lesbian youths: The role of internalized sexual stigma, self-disclosure, and individuals' sense of connectedness to the gay community. Addict Behav. 2010 Oct;35(10):896-9. doi: 10.1016/j.addbeh.2010.06.004. Epub 2010 Jun 11. PMID 20584573
- [Background] Eisenberg ME, Toumbourou JW, Catalano RF, Hemphill SA. Social norms in the development of adolescent substance use: a longitudinal analysis of the International Youth Development Study. J Youth Adolesc. 2014 Sep;43(9):1486-97. doi: 10.1007/s10964-014-0111-1. Epub 2014 Mar 15. PMID 24633850
- [Background] Mason TB, Lewis RJ, Gargurevich M, Kelley ML. Minority stress and intimate partner violence perpetration among lesbians: Negative affect, hazardous drinking, and intrusiveness as mediators. Psychology of Sexual Orientation and Gender Diversity. 2016;3(2):236-246.
- [Background] Edwards KM, Sylaska KM, Neal AM. Intimate partner violence among sexual minority populations: A critical review of the literature and agenda for future research. Psychology of Violence. 2015;5(2):112-121.
- [Background] Edwards KM, Sylaska KM. The perpetration of intimate partner violence among LGBTQ college youth: the role of minority stress. J Youth Adolesc. 2013 Nov;42(11):1721-31. doi: 10.1007/s10964-012-9880-6. Epub 2012 Dec 12. PMID 23233160
- [Background] Lewis RJ, Millentich RJ, Kelley ML, Woody A. Minority stress, substance use, and intimate partner violence among sexual minority women. Aggression and Violent Behavior. 2012;17:247-256.
- [Background] Kertzner RM, Meyer IH, Frost DM, Stirratt MJ. Social and psychological well-being in lesbians, gay men, and bisexuals: the effects of race, gender, age, and sexual identity. Am J Orthopsychiatry. 2009 Oct;79(4):500-10. doi: 10.1037/a0016848. PMID 20099941
- [Background] Lin Y, J., Israel T. Development and validation of a psychological sense of LGBT community scale. Journal of Community Psychology. 2012;40(5):14.
- [Background] Dank M, Lachman P, Zweig JM, Yahner J. Dating violence experiences of lesbian, gay, bisexual, and transgender youth. J Youth Adolesc. 2014 May;43(5):846-57. doi: 10.1007/s10964-013-9975-8. Epub 2013 Jul 17. PMID 23861097
- [Background] Noar SM, Pierce LB, Black HG. Can computer-mediated interventions change theortical mediators of safer sex? A meta-analysis. Human Communication Research. 2010;36:36.
- [Background] Bennett S, Banyard VL, Edwards KM. The Impact of the Bystander's Relationship With the Victim and the Perpetrator on Intent to Help in Situations Involving Sexual Violence. J Interpers Violence. 2017 Mar;32(5):682-702. doi: 10.1177/0886260515586373. Epub 2016 Jul 11. PMID 26037814
- [Background] Growing up LGBT in America: NCOD report. Human Rights Campaignn.
- [Background] GLSEN. The 2015 national school climate survey: Executive summary. GLSEN;2015.
- [Background] Lenhart A. A majority of American teens report access to a computer, game console, smartphone and a tablet. Washington, DC: Pew Research Center. 2015.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The PRYSHM program is theoretically grounded, follows best practices for effective health behavior prevention, and includes nine, one hour sessions co-facilitated by 2 LGBTQ+ adults.
- Waitlist Control: Check-ins/provision of resources
Period: Overall Study
Arm/Group | Intervention | Waitlist Control
Started | 213 | 101
Completed | 204 | 100
Not Completed | 9 | 1
Not completed — removed by researchers for offensive or deceptive behavior | 9 | 1

BASELINE CHARACTERISTICS:
Population: Of the 1662 individuals who sought consent, 1348 of them were either screened out or did not complete the survey. Therefore, 314 participants were then randomized into either intervention or waitlist control conditions. Of these 314 participants, ten (10) were removed by the researchers for offensive or deceptive behavior. Thus, the analysis population at baseline was 304.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Waitlist Control | Total
Number analyzed (Participants) | 204 | 100 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 204 | 100 | 304
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.53 (0.88) | 16.53 (0.9) | 16.53 (0.89)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Boy/Man | 32 | 15 | 47
  Girl/Woman | 66 | 30 | 96
  Trans | 1 | 0 | 1
  Genderqueer | 15 | 9 | 24
  Non-binary | 33 | 22 | 55
  Unsure/questioning | 7 | 1 | 8
  Other | 23 | 7 | 30
  Trans girl/woman | 1 | 1 | 2
  Trans boy/man | 25 | 14 | 39
  Refused | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 16 | 64
  Not Hispanic or Latino | 152 | 81 | 233
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 17 | 3 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 14 | 49
  White | 78 | 51 | 129
  More than one race | 59 | 25 | 84
  Unknown or Not Reported | 15 | 4 | 19
Region of Enrollment [Number; unit: participants]
  United States | 204 | 100 | 304

OUTCOME MEASURES:

1. Primary Outcome: Intimate Partner Violence Perpetration at Week 21
Description: The Measure of Adolescent Relationship Harassment and Abuse (MARSHA): Perpetration Scale assesses how often an individual perpetrates dating violence. Participants rate how frequently they engaged in specific behaviors from 0 to 100 times over the past three months (at Week 21). The total score was created by summing the items. The range is 0 to 476. Higher scores represent more intimate partner violence perpetration.
Time Frame: Week 21
Population: This number reflects the final number of participants in Week 21; 61 participants lost to attrition throughout the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 5.79 (39.85) | 4.46 (11.02)

2. Primary Outcome: Intimate Partner Violence Victimization at Week 21
Description: The Measure of Adolescent Relationship Harassment and Abuse (MARSHA): Victimization Scale assesses how often an individual experiences abusive behavior from a romantic partner. Participants indicate how often they have been the victim of abuse from 0 to 100 times in the past three months (at Baseline, Week 21). The total score was created by summing the items. The range is 0 to 105. Higher scores represent more intimate partner violence victimization.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
units on a scale | 5.57 (16.56) | 6.83 (19.73)

3. Primary Outcome: Alcohol Use at Week 21
Description: The Alcohol Use Questionnaire is based on the Daily Drinking Questionnaire and assesses an individual's alcohol use. Participants indicate how often they have used/abused alcohol within their lifetime, over the past 3 months on a scale of "0" to "40+". recoded the response scale using the mid-point of each response option (recoded values: 0 = 0, 1 = 1, 2 = 2, 3 = 3, 4 = 4, 5 = 5, 6 = 7.5, 7 = 14.5, 8 = 29.5, 9 = 40. Mean scores were then calculated. The range is 0 to 9. Higher scores represent more alcohol use.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.13 (2.58) | 1.86 (4.37)

4. Primary Outcome: Sexual and Gender Minority Specific Intimate Partner Violence Perpetration at Week 21
Description: The Conflict Tactics Scale-Revised: Sexual and Gender Minority Specific Intimate Partner Violence Perpetration (CTS-2:IPV-Perpetration, SGM specific) assesses how often an individual identifying as a sexual and/or gender minority perpetrates dating violence. Participants rate how frequently they engaged in specific behaviors from 0 to 100 times over the past three months (Week 21). The total score was created by summing the items. The range is 0 to 5. Higher scores represent more sexual and gender minority specific intimate partner violence perpetration.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
units on a scale | 0.04 (0.42) | 0.10 (0.54)

5. Primary Outcome: Sexual and Gender Minority Specific Intimate Partner Violence Victimization at Week 21
Description: The Conflict Tactics Scale-Revised: Sexual and Gender Minority Specific Intimate Partner Violence Victimization (CTS-2:IPV-Victimization, SGM specific) assesses how often an individual identifying as a sexual and/or gender minority victimizes dating violence. Participants rate how frequently they engaged in specific behaviors from 0 to 100 times over the past three months (Week 21). The total score was created by summing the items. The range is 0 to 16. Higher scores represent more sexual and gender minority specific intimate partner violence victimization.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
units on a scale | 0.35 (1.75) | 0.53 (1.91)

6. Primary Outcome: Drinking Intentions at Week 21
Description: The Drinking Intentions Questionnaire is an instrument based on the Daily Drinking Questionnaire and assesses how likely an individual is to drink in the future. Participants to rate how likely they are to drink alcohol in the next three months (Week 21) on a scale of 0 to 4 ("definitely will" to "definitely won't") on one item. The range is 0 to 4. Higher scores represent more drinking intentions.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.50 (1.35) | 1.32 (1.33)

7. Primary Outcome: Willingness to Drink at Week 21
Description: The Willingness to Drink Questionnaire assesses intensity of drinking behavior. Participants rate how likely they would be to drink at varying levels of intensity on a scale from 0 to 3 ("not at all" to "very willing") given a specific scenario. The mean score was created. The range is 0 to 3. Higher scores represent more willingness to drink
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.20 (1.00) | 1.04 (0.98)

8. Secondary Outcome: Experience of Negative Consequences as a Result of Alcohol Use at Week 21
Description: The Brief Young Adult Alcohol Consequences Questionnaire is a validated, self-report instrument assessing the frequency with which an individual has experienced negative consequences as a result of drinking alcohol. Participants are asked to indicate if they have experienced a specific consequence of drinking alcohol in the past three months (Week 21) with a "yes" or "no" answer. The number of "yes" responses provides an indication of the severity of alcohol-related consequences. The total score was created by summing the items. The range is 0 to 24. Higher scores represent higher levels of problems and consequences from alcohol use.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.01 (2.71) | 1.26 (2.94)

9. Secondary Outcome: Depressive Symptoms at Week 21
Description: The construct will be measured using 8 items from the Patient Health Questionnaire-9 Item (PHQ-9) which is a validated, self-report instrument assessing experience of symptoms associated with major depressive disorder. Participants are asked to measure how many days in the past two weeks they have experienced a symptom of depression on a scale of 0 (not at all) to 3 (nearly every day). The sum of all responses is used to indicate likelihood of major depressive disorder. Higher scores indicate higher depressive symptomology.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 9.07 (6.35) | 10.00 (5.90)

10. Secondary Outcome: Drug Use at Week 21
Description: The construct will be measured using two questions from the Youth Risk Behavior Surveillance (YRBS) questionnaire that address drug use. Participants are asked to indicate if they have used specific drugs in the past three months (Week 21) with either 1) yes or 0) no. The range is 0 to 1. A score of 1 indicates the use of drugs and therefore is considered a worse outcome.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 0.38 (0.49) | 0.44 (0.50)

11. Secondary Outcome: Sexual Risk-Taking as Measured by the Sexual Risk Survey at Week 21
Description: The Sexual Risk Survey is a validated self-report measure assess how often an individual has engaged in risky sexual behavior. Participants indicate how often they have engaged in risky sexual behaviors in the past three months (week 21) on a scale of "0" to "30+". A composite score was created by recoding each item (0, 1, and 2 or more) and then creating a sum. The range is 0 to 8. Higher scores indicate higher levels of sexual risk.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 2.13 (2.17) | 1.82 (2.03)

12. Other Pre Specified Outcome: Identity Concealment Behaviors as Measured by the Outness Inventory for Sexual Orientation Family Subscale at Week 21
Description: The Outness Inventory for Sexual Orientation Family Subscale is a modified measures that determine to what extent an individual's family members knows about the sexual orientation of the individual. Scores are analyzed as a sum of individuals and groups who are aware of the individual's sexual orientation. The range is 0 to 1. Higher scores indicate higher levels of outness.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 0.89 (0.29) | 0.92 (0.27)

13. Other Pre Specified Outcome: Experiences of Internalized Homonegativity at Week 21
Description: The Adapted Homonegativity Items constitute a validated self-report measure that assesses to what extent an individual experiences internalized homonegativity. Individuals are asked to indicate their agreement with specific statements representing internalized homonegativity on a scale from 1 (strongly disagree) to 4 (strongly agree). Responses are averaged to provide an indication of internalized homonegativity. The range is 1 to 4. Higher scores indicate higher levels of internalized stigma.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.83 (0.61) | 1.97 (0.69)

14. Other Pre Specified Outcome: Sense of LGBTQIA2S+ Community at Week 21
Description: The Psychological Sense of LGBT Community is a validated, self-report measure that assesses the extent to which an individual feels they belong to and contribute to the LGBTQIA2S+ community. Participants rate how often they feel specific indicators of LGBTQIA25+ community on a scale from 1 (none) to 5 (a great deal). The measure provides two subscales: needs fulfillment and membership. Responses within each subscale and overall scale are calculated to provide a mean score. Higher scores indicate higher levels of sense of community.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale
  Membership Subscale | 3.25 (0.90) | 2.96 (1.14)
  Needs Fulfilment | 2.80 (0.89) | 2.59 (0.99)

15. Other Pre Specified Outcome: Emotional Regulation and Coping at Week 21
Description: The Difficulties in Emotion Regulation Scale (DERS-16): Impulse Control Subscale assesses an individual's capacity for impulse control. Participants rate how often they feel out of control of their emotions when upset on a scale of 1 (almost never) to 5 (almost always). Responses are summed with higher scores reflecting greater levels of emotional dysregulation. The range is 3 to 15.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 6.77 (2.91) | 6.40 (2.97)

16. Other Pre Specified Outcome: Conflict Resolution Skills as Measured by the Communication Skills Test at Week 21
Description: The Communication Skills Test: 10-Item Version (CST-10) is a validated, self-report measure which assesses how likely an individual is to utilize specific conflict resolution skills when experiencing conflict with a romantic partner. Participants are asked to rate how easy or difficult it would be to engage in specified de-escalation strategies on a scale of 1 (very difficult) to 4 (very easy). The scale is computed by creating a mean score from the item responses, including reverse-scored items. The range is 1 to 4. Higher scores indicate higher levels of conflict resolution skill self-efficacy.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 3.21 (0.51) | 3.20 (0.49)

17. Other Pre Specified Outcome: Sexual Refusal Skills at Week 21
Description: The Sexual Communication Self-Efficacy Scale assesses capacity for refusal during intimate interactions. Participants rate how difficult it would be to refuse a sexual request on a scale of 1 (very difficult) to 4 (very easy). The measure provides two subscales: negative sexual messages, positive sexual messages. The respective subscale scores are calculated by taking the means of the subscale's items. The range is 1 to 4. Higher scores indicate higher levels of sexual communication self-efficacy.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale
  Negative messages | 3.14 (0.72) | 3.16 (0.73)
  Positive Messages | 3.13 (0.71) | 3.22 (0.73)

18. Other Pre Specified Outcome: Bystander Behavior at Week 21
Description: Bringing in the Bystander Intervention Items assesses the capacity to intervene in instances of dating violence. Participants rate how likely they would be to intervene in a specific situation from 1 to 4 ("very unlikely" to "very likely"). The measure provides two subscales: reactive and proactive. Subscale scores are calculated by summing item responses and then dividing by the number of items to produce a mean subscale score. The summed ranges are 6 to 24 for reactive subscale with 6 items. The summed ranges are 3 to 12 for proactive subscale with 3 items. Higher scores indicate higher levels of bystander behavior intentions on each of the two subscales.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale
  Reactive | 3.58 (0.43) | 3.51 (0.52)
  Proactive | 3.49 (0.59) | 3.46 (0.67)

19. Other Pre Specified Outcome: Accurate Perceptions of Dating Violence at Week 21
Description: The Perceived Dating Violence Norms, adapted from the Measure of Adolescent Relationship Harassment and Abuse (MARSHA)-Perpetration scale, assesses an perceptions of dating violence within LGBTQIA2S+ teenage relationships. Participants indicate what percentage of LGBTQIA2S+ teenage relationships they believe experience specific scenarios related to abuse. The measure provides 6 subscales: social control, physical abuse, sexual abuse, isolation, cyber control, intimidation. Subscale scores are calculated by averaging item responses on the respective subscale. The range is 0 to 73.81. Higher scores represent more perceived dating violence norms.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 13.36 (15.03) | 16.39 (15.87)

20. Other Pre Specified Outcome: Protective Behavioral Strategies as Measured by the Alcohol Reduction Strategies- Current Confidence Questionnaire (ARS-CC) at Week 21
Description: The Alcohol Reduction Strategies- Current Confidence Questionnaire (ARS-CC) is a validated, self-report measure which assesses an individual's use of alcohol reduction strategies to prevent negative consequences associated with alcohol use. Participants are asked to rate how confident they are in their ability to utilize a given strategy on a 5 point scale of 1 (not at all confident) to 5 (completely confident). Responses are averaged to provide an overall mean score, with a higher indicating a greater capacity to utilize alcohol reduction strategies.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 4.04 (0.83) | 3.88 (0.87)

21. Other Pre Specified Outcome: Hope for the Future as Measured by the Feelings About Being LGBTQIA2S+ at Week 21
Description: The Feelings about Being LGBTQIA2S+ is a validated, self-report measure which assesses an individual's feelings toward the future as an LBGTQIA2S+ individual. Participants are asked to rate the likelihood of experiencing positive life outcomes as an LBGTQIA2S+ individual on a scale of 1 (definitely no) to 4 (definitely yes). Response items are averaged to provide an overall score, with higher scores indicating a more positive outlook. The range is 1 to 4.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 3.34 (0.55) | 3.25 (0.68)

22. Other Pre Specified Outcome: Drinking Motives at Week 21
Description: The Drinking Motives Questionnaire- Revised (DMQ-R) assesses the extent to which a participant uses alcohol to cope with negative emotions. Participants indicate how often they experience a given motive for drinking on a scale of 0 (almost never/never) to 5 (almost always/always). Scale scores are calculated as the sum of the respective items, with higher scores indicating a greater likelihood that a participant uses alcohol to cope with negative emotions. The range is 0 to 5.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.02 (0.89) | 1.04 (1.11)

23. Other Pre Specified Outcome: Drinking Refusal Skills at Week 21
Description: The Drinking Refusal Self-Efficacy Questionnaire- Shortened Adolescent Version (DRSEQ-SRA) assesses individual capacity to resist alcohol use. Given a scenario, participants rate their ability to refuse alcohol from "I am very sure I could NOT resist drinking" to "I am very sure I could resist drinking". Two subscales are provided: social pressure, emotional relief. Total and subscale scores are calculated by summing item responses on the total measure and respective subscales. The range for both social pressure and emotional relief subscales is 6 to 36. Higher scores in both subscales indicate higher levels of drinking refusal self-efficacy. Higher scores indicate higher levels of drinking refusal self-efficacy.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale
  Social pressure | 14.63 (3.84) | 14.42 (4.05)
  Emotional relief | 15.88 (3.59) | 16.25 (3.20)

24. Other Pre Specified Outcome: Alcohol Use Bystander Behavior at Week 21
Description: The Alcohol Use: Likelihood to Intervene assesses the capacity to intervene in situations of alcohol abuse and addiction. Participants are asked to rate how likely they would be to intervene in specific situations on a scale of 1 (very unlikely) to 4 (very likely). Responses across items are averaged to provide an overall score, with a higher score indicating a greater capacity to intervene. The range is 1 to 4.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 3.66 (0.55) | 3.63 (0.46)

25. Other Pre Specified Outcome: Accurate Perceptions of Alcohol Use at Week 21
Description: The Drinking Norms Rating Form, adjusted to LGBTQIA2S+ populations, assesses an individual's perception of drinking behavior of LGBTQIA2S+ teens. Participants indicate what percentage of LGBTQIA2S+ teens they believe engage in specific drinking behaviors. Percentages are averaged to indicate perception ranging from 0 = 0 times to 9 = 40+ times. We recoded the response scale using the mid-point of the response options. The range is 0 to 40. Higher scores represent higher levels of perception of social norms.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 4.48 (6.79) | 6.04 (8.05)

26. Other Pre Specified Outcome: Ethnic Identity at Week 21
Description: The Multi-Group Ethnic Identity Measure assesses adolescents' perceived affirmation and sense of belonging to their ethnic identity. Participants indicate how much they agree on a five point scale with each of 13 statements about their ethnic identity. Mean scores were created for each subscale and higher scores represented higher levels of cognitive clarity, affective pride, or behavioral engagement. The ranges are all from 1 to 5.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale
  Cognitive clarity | 3.47 (0.84) | 3.27 (1.09)
  Affective pride | 3.63 (0.94) | 3.38 (1.19)
  Behavioral engagement | 3.32 (0.88) | 3.02 (1.07)

27. Other Pre Specified Outcome: Identity Concealment Behaviors as Measured by the Outness Inventory for Sexual Orientation World Subscale at Week 21
Description: The Outness Inventory for Sexual Orientation World Subscale is a modified measures that determine to what extent an individual's social network knows about the sexual orientation of the individual. Scores are analyzed as a sum of individuals and groups who are aware of the individual's sexual orientation. The range is 0 to 4. Higher scores indicate higher levels of outness.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.86 (0.83) | 1.79 (0.90)

28. Other Pre Specified Outcome: Identity Concealment Behaviors as Measured by the Outness Inventory for Gender Identity Family Subscale at Week 21
Description: The Outness Inventory for Gender Identity Family Subscale is a modified measure that determine to what extent an individual's family members know about the gender identity of the individual. A summed total composite score was used to create a mean average score. The range is 0 to 1. Higher scores indicate higher levels of outness.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 0.89 (0.32) | 0.77 (0.38)

29. Other Pre Specified Outcome: Identity Concealment Behaviors as Measured by the Outness Inventory for Gender Identity World Subscale at Week 21
Description: The Outness Inventory for Gender Identity Family Subscale is a modified measures that determine to what extent an individual's social networks knows about the gender identity of the individual. Scores are analyzed as a sum of individuals and groups who are aware of the individual's gender identity. The range is 0 to 4. Higher scores indicate higher levels of outness.
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 170 | 83
score on a scale | 1.87 (1.10) | 1.82 (1.10)

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected throughout the study from baseline (enrollment 1-2 weeks before programming), during intervention (9-week programming), post-program survey (within 3 weeks of program end), 3-month follow-up from baseline, and during waitlist control intervention programming (at month 12 (9-weeks of programming)).
Description: All-Cause Mortality is not a possible outcome of this trial.
Groups:
- Waitlist Control: Treatment Condition: Received PRYSHM program intervention following the completion of ALL data collection.
Arm/Group | Treatment Condition | Waitlist Control | Waitlist Control: Treatment Condition
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/100 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/100 | 0/16
Other Adverse Events (participants affected / at risk) | 6/204 | 0/100 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Condition (N=204) | Waitlist Control (N=100) | Waitlist Control: Treatment Condition (N=16)
Other (Not Including Serious) Adverse Events (Social circumstances) | 6 (6) | 0 (0) | 0 (0) — During a program session, a participant spontaneously displayed a hate symbol that other participants saw; participants reported being upset by the hate symbol.
Other (Not Including Serious) Adverse Events (Social circumstances) | 1 (1) | 0 (0) | 0 (0) — A student researcher meant to email the PI but accidentally emailed someone with a similar name. The email contained the name of a participant but no other information. The email was deleted by the person who received it in error right away.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05521906/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05521906/SAP_002.pdf
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05521906/ICF_000.pdf